CLINICAL TRIAL: NCT03176524
Title: A Randomised, Double-blind, Three-period Crossover Trial to Investigate the Safety and the Pharmacokinetic, Pharmacodynamic Characteristics of Two BioChaperone® Glucagon Formulations Compared to Marketed GlucaGen® in Subjects With Type 1 Diabetes
Brief Title: A Trial to Investigate the Safety and the Pharmacokinetic, Pharmacodynamic Characteristics of Two BioChaperone® Glucagon Formulations Compared to Marketed GlucaGen® in Subjects With T1DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC13-CT028
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BioChaperone® glucagon formulation 1 (Experimental): Single subcutaneous fixed doses (50 µg and 1.0 mg)
  Interventions: Drug: BioChaperone® glucagon formulation 1
- BioChaperone® glucagon formulation 2 (Experimental): Single subcutaneous fixed doses (50 µg and 1.0 mg)
  Interventions: Drug: BioChaperone® glucagon formulation 2
- GlucaGen® HypoKit® (Active Comparator): Single subcutaneous fixed doses (50 µg and 1.0 mg)
  Interventions: Drug: GlucaGen® HypoKit®

INTERVENTIONS:
Drug: BioChaperone® glucagon formulation 1 — Injection of BioChaperone® glucagon formulation 1 at Day 1: 50 µg and at Day 2: 1 mg
  Arms: BioChaperone® glucagon formulation 1
Drug: BioChaperone® glucagon formulation 2 — Injection of BioChaperone® glucagon formulation 2 at Day 1: 50 µg and at Day 2: 1 mg
  Arms: BioChaperone® glucagon formulation 2
Drug: GlucaGen® HypoKit® — Injection of GlucaGen® HypoKit® at Day 1: 50 µg and at Day 2: 1 mg
  Arms: GlucaGen® HypoKit®

SUMMARY:
This is a single centre, double-blind, randomised, three-period crossover phase 1 trial in subjects with type 1 diabetes mellitus (T1DM). Each subject will be randomly allocated to a sequence of three treatments, i.e. two single subcutaneous doses of BioChaperone® Glucagon (BC Glucagon) formulation 1, BioChaperone® Glucagon formulation 2 and GlucaGen® HypoKit®, each at the fixed doses of 50 µg and 1 mg on 3 separate dosing visits.

Following trial drug administration, pharmacokinetics (PK) and pharmacodynamics (PD) assessments will be carried until 4 hours. Safety will be assessed during all the trial period.

The total trial maximum duration for the individual subject will be up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 64 years (both inclusive)
* Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months prior to the screening visit
* Treated with daily insulin for T1DM ≥ 12 months prior to the screening visit
* Stable insulin treatment at least 3 months prior to the screening visit
* Stable disease with HbA1c <9.0 %
* C peptide <=0.30 nmol/L
* Body mass index (BMI) < 30.0 kg/m2

Exclusion Criteria:

* Type 2 Diabetes mellitus
* Previous participation in this trial. Participation is defined as being randomised
* Receipt of any medicinal product in clinical development within 60 days prior to this trial
* Clinically significant abnormal haematology, biochemistry, urinalysis, or coagulation screening tests, as judged by the Investigator considering the underlying disease
* Known or suspected hypersensitivity to the trial products or related products
* Severe hypoglycaemic events within one month prior to screening, as judged by the investigator
* Recent administration of glucagon (within 3 months prior to Screening)
* Clinically relevant diabetic complications as judged by the investigator
* Women of child bearing potential not willing to use contraceptive methods

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Clinical safety laboratory | Up to 10 weeks
  Haematology, biochemistry and urinalysis: changes or findings from baseline in clinical safety laboratory parameters during the trial duration (screening visit, treatment visits and follow up visit)
Physical examination | Up to 10 weeks
  Examination of the body systems
ECG parameters | Up to 10 weeks
  Heart rate, PQ, QRS, QT, QTcB: changes or findings from baseline in ECG parameters during the trial duration (screening visit, treatment visits and follow up visit)
Vital signs | Up to 10 weeks
  Diastolic and systolic blood pressure (mmHg), Pulse (beats/min), Body temperature (°C), Respiratory frequency (RF/min): changes or findings from baseline in vital signs during the trial duration (screening visit, treatment visits and follow up visit)
Adverse events and serious adverse events | Up to 10 weeks
  Untoward medical occurrence
Assessments of local tolerability at injection site | Up to 10 weeks
  Local reaction at injection site

SECONDARY OUTCOMES:
AUCPK 0-30min | From 0 to 30 min
  area under the baseline adjusted plasma glucagon concentration curve from 0 to 30 min
AUC PK 0-4h | From 0 to 4 hours
  area under the baseline adjusted plasma glucagon concentration curve from 0 to 4 h
ΔAUCPG 0-30min | From 0 to 30 min
  area under the baseline adjusted plasma glucose curve from 0 until 30 min
ΔAUCPG 0-4h | From 0 to 4 hours
  area under the baseline adjusted plasma glucose curve from 0 until 4h
ΔPG 30min | From 0 to 30 min
  baseline adjusted plasma glucose concentration at 30 min
Percentage of patients achieving a plasma glucose increase of ≥20 mg/dL from baseline within 30 minutes after treatment | 30 min after drug administration
  only at day 2
Time to plasma glucose increase of ≥20 mg/dL from baseline | Up to 4 hours after drug administration
  only at day 2

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No